CLINICAL TRIAL: NCT01086163
Title: Effects of Prescription OMega-3 Fatty Acids (Omacor®, Lovaza®) on Platelet Activity in Patients With Coronary Artery Disease With Hypertriglyceridemia (OMPA-CAD)
Brief Title: Effects of Omega-3 Fatty Acids on Platelets in Patients With Coronary Artery Disease With Hypertriglyceridemia
Acronym: OMPA-CAD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HeartDrug Research LLC (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Dr. Victor Serebruany. MD, PhD, HeartDrug Research laboratories
Other Study IDs: HD-Oma-09/27D
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Coronary Artery Disease
Keywords: Omacor; Simvastatin; Aspirin; Platelet activity; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Omacor; Fatty Acids, Omega-3

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serial blood samples - at baseline, day 7, and day 14 after treatment assignment
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Omacor dose titration: Stable documented coronary artery disease proven by angiography treated with statin and aspirin. In order to achieve homogeneity within this population, the following additional inclusion criteria will apply:
  * survived first-time AMI more than 12 months ago
  * stable medical treatment during the last 3 months (except removal of Plavix)
  * Ethnicity: Caucasians
  * Males, 50 - 60 yrs
  * non-diabetics
  * excluded are those who eat more than one meal of fish / week
  * excluded are those who take omega-3 supplements of any sorts
  Interventions: Drug: Omacor, omega-3 fatty acids in CAD patients

INTERVENTIONS:
Drug: Omacor, omega-3 fatty acids in CAD patients — Omacor 1g versus 2g daily versus placebo
  Other Names: Lovaza

SUMMARY:
Omacor®/Lovaza® is an effective, and very safe mix of PO-3A, and the drug is currently approved by the Federal authorities for the drug management of post-infarction patients with high blood triglycerides. Given the growing length of CAD progression, it is pertinent that many more patients will yield extra benefit from Lovaza® on top of aggressive antiplatelet regimens and statin due to severity of their vascular disease. Therefore, mild antiplatelet properties of PO-3A will be a highly desirable and attractive commodity of this medication.

The investigators believe that Omacor®/Lovaza® is ideally positioned for the chronic management of CAD as a safe, efficient, and "gentle" agent with no harmful interactions with statins or aspirin.

The investigators hypothesize that addition of Omacor may add mild antiplatelet protection for CAD patients.

The study objectives are:

* To assess the ex vivo effects of Omacor® on platelet function in patients with coronary artery disease (CAD).
* To compare ex vivo platelet-related effects after 7 and 14 days of therapy with Omacor and statin combination versus statin alone in patients with chronic stable coronary heart disease.
* To establish the relation of changes in platelet activity (if any) with the lipid profile to prove an additional benefit of Omacor® on top of statin and aspirin.

DETAILED DESCRIPTION:
In terms of incidence, prevalence, morbidity, and economic costs, coronary artery disease represents a number 1 public health concern. Omacor®/Lovaza® is an effective, and very safe mix of PO-3A, and the drug is currently approved by the Federal authorities for the drug management of post-infarction patients with high blood triglycerides. Despite significant progress in the prevention and treatment of vascular disease in the Western World in the past two decades, national statistics indicate that the incidence and prevalence of heart disease has been increasing steadily. Given the growing length of CAD progression, it is pertinent that many more patients will yield extra benefit from Lovaza® on top of aggressive antiplatelet regimens and statin due to severity of their vascular disease. Therefore, mild antiplatelet properties of PO-3A will be a highly desirable and attractive commodity of this medication.

We believe that Omacor®/Lovaza® is ideally positioned for the chronic management of CAD as a safe, efficient, and "gentle" agent with no harmful interactions with statins or aspirin. Also considering low clinical incidence of aspirin-induced interactions with other classes of drugs, Lovaza® may fit nicely into a standard cocktail for diabetes, hypertension, depression, arrhythmias, and heart failure management of CAD patients, which will expand the drug utilization. However, platelet-related effects of Lovaza® on top of aspirin and statin in patients with stable coronary disease are not known, but may be important due to the high incidence of aspirin resistance and heavy burden of thrombin activation in such patients. We have a large pool of patients with documented CAD (300-350/annum), and we will be able to enroll relatively large amount of quality patients fast.

ELIGIBILITY:
Inclusion Criteria:

* Stable documented coronary artery disease proven by angiography treated with statin and aspirin. In order to achieve homogeneity within this population, the following additional inclusion criteria will apply:
* survived first-time AMI more than 12 mths ago
* stable medical treatment during the last 3 months (except removal of Plavix)
* Ethnicity: Caucasians
* Males, 50 - 60 yrs
* Non-diabetics
* Excluded are those who eat more than one meal of fish / week
* Excluded are those who take omega-3 supplements of any sorts

Exclusion Criteria:

* Thrombolytic therapy or GP IIb/IIIa inhibitor within 30 days of enrollment
* Platelet count < 100,000
* History of bleeding disorder
* Hct < 30, serum creatinine ≥3 mg/dL, liver impairment defined as ALT/AST > 3 times upper limit of normal.
* Glomerular filtration rate <50ml/min
* Admission for acute vascular syndrome (unstable angina, MI, stroke), revascularization procedure with stent placement, or other major coronary/cerebrovascular event within 30 days.
* Active participation in other investigational drug or device trial within the last 30 days.
* Allergy or intolerance to any of the study medications.
* Antiplatelet agent other than aspirin or
* Insulin therapy
* Cancer of any localization

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Serial assessments of platelet characteristics from 10 patients in each of the 3 study groups at 2 time points for the total of 60 platelet samples. First, patients with stable coronary disease will be identified, telephone interviews will be conducted, and screening visits scheduled to those who qualify. We expect to triage 50 patients who then will be examined, and biochemistry markers tested. Patients will be allocated to one of three treatment arms based on randomization. Enrollment will continue until all 3 cells will be filled (n=10 each).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-02 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Change in platelet aggregation after Lovaza® (1 or 2g/daily) in patients treated with aspirin + simvastatin versus those matched patients treated with placebo+aspirin +simvastatin in combination. | Day 7 and Day 14

SECONDARY OUTCOMES:
Differences in expression of P-selectin and PAR-1 receptors after treatment with Lovaza® (1 or 2g/daily) in patients treated with aspirin + simvastatin versus those matched patients treated with placebo+aspirin +simvastatin in combination. | Day 7 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Alex Pokov, MD, Study Chair — HeartDrug Research
Locations (1):
- Victor Serebruany, Towson, Maryland, United States